CLINICAL TRIAL: NCT01775410
Title: A Non-randomized, Multi-center Feasibility Trial of the Avinger Wolverine System, an Atherectomy Device That Provides Directional Visualization and Imaging While Removing Plaque in Diseased Lower Extremity Arteries
Brief Title: OptiCal COherence ToMography ABoard InformiNg AtherEctomy
Acronym: COMBINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was terminated by sponsor without any AEs to review the device design.
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P 0218
Record Dates: First submitted 2013-01-14; First posted 2013-01-25 (Estimated); Results first posted 2021-04-21 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2021-04

CONDITIONS: Atherectomy in Diseased Lower Extremity Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Wolverine System (Experimental): Wolverine System to perform atherectomy while using directional visualization and imaging as an adjunct to fluoroscopy to aid removal of plaque from diseased lower extremity arteries
  Interventions: Device: Wolverine System to perform atherectomy

INTERVENTIONS:
Device: Wolverine System to perform atherectomy

SUMMARY:
This is a prospective, multi-center, non-randomized single arm feasibility trial of the Wolverine OCT guided atherectomy system.The trial will enroll up to 50 subjects diagnosed with peripheral vascular disease of the lower extremities.The primary disease must be located in reference vessel diameters ≥ 2.5 mm which is significant enough to cause moderate to severe symptoms and warrant vascular intervention.

DETAILED DESCRIPTION:
This is a prospective, multi-center, non-randomized single arm feasibility trial of the Wolverine OCT guided atherectomy system. The trial is predominantly descriptive and, as such, not powered statistically although endpoint comparisons may be made to the published literature on peripheral atherectomy.

The trial will enroll up to 50 subjects diagnosed with peripheral vascular disease of the lower extremities. The primary disease must be located in reference vessel diameters ≥ 3.0 mm which is significant enough to cause moderate to severe symptoms and warrant vascular intervention. Trial success is focused on short term safety including rates of major adverse events. An evaluation of efficacy will also be performed and will include an evaluation of technical success defined as the percent of target lesions that has a residual diameter stenosis <50% post the Wolverine device alone as assessed by an independent review at the time of treatment using quantitative angiography or visual estimate.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Patient is a candidate for percutaneous intervention for peripheral vascular disease in the legs.
3. Patient is willing and able to give informed consent
4. Documented symptomatic atherosclerotic peripheral vascular disease Rutherford Classification 2-5.
5. Reference vessel lumen proximal to target lesion >2.5 mm in diameter by visual estimation.
6. Subject has de novo target lesion(s) with stenosis >70% by visual estimation distal to the profunda femoral artery. No more than 2 lesions may be treated with the Wolverine device.
7. Target lesion length <10 cm if target lesion >70% and <99% stenosed. If target lesion a chronic total occlusion (99-100% stenosed), target lesion length <4 cm.
8. Patient is capable of meeting requirements and be present at the follow-up clinic visits at 30 days.
9. At least one patent tibial run-off vessel at baseline.

Exclusion Criteria:

1. Subject is pregnant or breast feeding.
2. Rutherford Class 0 to 1 (asymptomatic and mild claudication).
3. Rutherford Class 6 (critical limb ischemia).
4. Severe calcification of the target lesion.
5. Target lesion with any type of stent or graft.
6. Target lesion in the iliac artery.
7. Target lesion stenosis <70%.
8. Subjects with significant (>70%) occlusive lesions proximal to the target lesion not successfully treated during the index procedure (upstream disease) and prior to treatment of the target lesion.
9. Endovascular or surgical procedure performed on the index limb less than or equal to 30 days prior to the index procedure.
10. Planned endovascular or surgical procedure 30 days after the index procedure.
11. Lesion in the contralateral limb requiring intervention during the index procedure or within 30 days of the index procedure.
12. Subjects with active infections whether they are being currently treated or not.
13. Hemodialysis or GFR <30 mL/min or creatinine level >2.5mg/dL.
14. Evidence or history of intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stroke within the past 2 months.
15. Evidence or history of aneurysmal target vessel within the past 2 months.
16. History of severe trauma, fracture, major surgery or biopsy of a parenchymal organ within the past 14 days.
17. Known allergy to contrast agents or medications used to perform endovascular intervention that cannot be adequately pre-treated.
18. Subjects in whom anti-platelet, anticoagulant, or thrombolytic therapy is contraindicated.
19. History of heparin-induced thrombocytopenia (HIT).
20. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count less than 125,000/mm2 , known coagulopathy, or INR >1.5.
21. Any thrombolytic therapy within 2 weeks of the index procedure.
22. Any clinical and/or angiographic complication attributed to the use of another device prior to the insertion of the Wolverine into the subject.
23. Subjects or their legal guardians who have not or will not sign the Informed Consent.
24. Subjects who are unwilling or unable to comply with the follow-up study requirements.
25. Participation in any study of an investigational device, medication, biologic or other agent within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John B Simpson, MD, Study Director — Avinger, Inc.
Locations (2):
- Colombia (2):
  - Angiografia de Occidente, Cali, VAC
  - Clinical Cardiovascular, Medellín

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Wolverine System
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Colombia | 4
Target lesion length in cm [Mean (Standard Deviation); unit: cm] | 8.5 (1.7)
Vessel Luminal diameter in cm [Mean (Standard Deviation); unit: cm] | 3.8 (0.65)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With no Major Adverse Events
Description: Freedom from major adverse events (MAE) through 30 day follow-up:
  * Clinically driven target lesion revascularization (TLR)
  * Myocardial infarct (MI)
  * Cardiovascular related deaths
  * Unplanned, major index limb amputation
  * Device Related Events:
    * Clinically Significant Perforations
    * Clinically Significant Dissections
    * Clinically Significant Embolus
    * Pseudoaneurysm
Time Frame: Through 30 day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
Participants | 4

2. Secondary Outcome: Technical Success: Percent of Target Lesions That Have a Residual Diameter Stenosis < 50%
Description: Technical success is defined as the percent of target lesions that has a residual diameter stenosis < 50% post the Wolverine device alone as assessed by an independent review at the time of treatment using quantitative angiography or visual estimate
Time Frame: During interventional procedure
Measure: Number; unit: Percentage of target lesions
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
Percentage of target lesions | 100

3. Secondary Outcome: Procedural Success: Percent of Target Lesions That Have Residual Diameter Stenosis ≤30% Post-Wolverine and Any Other Adjunctive Therapy
Time Frame: Day 0
Measure: Number; unit: Percentage of target lesions
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
Percentage of target lesions | 100

4. Secondary Outcome: Number of Participants With no Procedural Emboli
Description: A procedural emboli is defined as a new occlusion of any visualized runoff vessel which cannot be reversed with an intravascular vasodilator.
Time Frame: During interventional procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
Participants | 4

5. Secondary Outcome: Ankle-Brachial Index (ABI) at 30 Days
Description: Ankle-Brachial Index (ABI) is the ratio of blood pressure in the lower legs to the blood pressure in the arms. It is calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressure in the arm.
  ABI < 0.95 indicates arterial disease; ABI between 0.95 and 1.3 is considered normal (free from significant peripheral artery disease); ABI > 1.3 is abnormal, and suggests calcification of the artery walls and incompressible vessels, indicating severe peripheral vascular disease.
Time Frame: At 30 days
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
Ratio | 1.32 (0.85)

6. Secondary Outcome: Rutherford Classification at 30 Days Post-procedure
Description: Rutherford Classification is a commonly used clinical means for describing the degree of peripheral artery disease. Rutherford Classifications range from Class 0: Asymptomatic, to Class 6: Major Tissue Loss. A lower score is less severe disease and a higher score is more severe disease progression.
Time Frame: At 30 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wolverine System
Number analyzed (Participants) | 4
score on a scale | 2.6 (0.63)

ADVERSE EVENTS:
Arm/Group | Wolverine System
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wolverine System (N=4)
Dissection (Vascular disorders) | 2 (2) — Dissection of the vessel wall

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less